CLINICAL TRIAL: NCT02386852
Title: Ginseng and Ginkgo Biloba Effects on Cognition as Modulated by Cardiovascular Reactivity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sunway University (Other)
Responsible Party: Principal Investigator, Dr. Luca Aquili, Dr. Luca Aquili, Sunway University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Sunway-979
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Blood Pressure; Cognition
Keywords: Ginseng; Ginkgo Biloba; cardiovascular reactivity; cognition
MeSH Terms: interventions — Asian ginseng; Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Experimental): Study subjects received, in a double blind fashion, placebo pills identical to the drug (ginseng: group 1; ginkgo biloba: group 2).
  Interventions: Drug: Placebo; Drug: Ginseng; Drug: Ginkgo Biloba
- Ginseng (Experimental): Participants in the ginseng group received a medium, and higher dose of ginseng in addition to placebo capsules.
  Interventions: Drug: Placebo; Drug: Ginseng
- Ginkgo Biloba (Experimental): Participants in the ginkgo biloba group received a medium, and higher dose of ginkgo in addition to placebo capsules.
  Interventions: Drug: Placebo; Drug: Ginkgo Biloba

INTERVENTIONS:
Drug: Placebo — Study subjects received, in a double blind fashion, placebo pills identical to the drug (drug 1-ginseng, group 1; drug 2-ginkgo biloba-group 2)
Drug: Ginseng — The ginseng group received two capsules containing either 1000 mg or 500 mg of Panax Ginseng extract standardized to 3% of ginsenosides (GNC, USA) or similarly looking placebo capsules over a period of three days of testing.
  Arms: Ginseng; Placebo
Drug: Ginkgo Biloba — The ginkgo group received two capsules containing either 240 mg or 120 mg of ginkgo biloba extract standardized to 24% ginkgo flavone glycosides and 6% terpene lactones (GBE24/6) or similarly looking placebo capsules over a period of three testing days.
  Arms: Ginkgo Biloba; Placebo

SUMMARY:
There is some evidence to suggest that ginseng and Ginkgo biloba can improve cognitive performance, however, very little is known about the mechanisms associated with such improvement. Here, we tested whether cardiovascular reactivity to a task is associated with cognitive improvement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ranging in age between 18 and 30.

Exclusion Criteria:

* Ginseng group: exclude those that regularly consume caffeine or Panax Ginseng, or those that are diabetic, have hormone sensitive conditions, autoimmune diseases, bleeding conditions, heart conditions or take medications that are known to interact with Panax Ginseng. These include anticoagulants, Warfarin, Ibuprofen, MAOIs, medications that are changed by the liver, and stimulant drugs (e.g. pseudoephedrine, epinephrine).
* Ginkgo Biloba group: exclude those that regularly consume caffeine or Ginkgo Biloba, or those that are diabetic, have experienced seizures in the past, have bleeding disorders, or take medications that are known to interact with Ginkgo Biloba. These include Ibuprofen, anticoagulants, Warfarin, Buspirone, Fluoxetine, Trazodone

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Cognitive performance as modulated by either ginseng or ginkgo biloba | Acute effects (3 days of testing)
  Cognitive effects on tests of vigilance/attention, behavioural flexibility and executive functioning

SECONDARY OUTCOMES:
Cardiovascular reactivity as a result of ginseng or ginkgo biloba intake | Acute effects (3 days of testing)
  Changes in systolic, diastolic and heart rate reading as a result of ginseng or ginkgo biloba intake and dependent upon the type of cognitive domain assessed (i.e. vigilance, behavioural flexibility or executive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Aquili, PhD, Principal Investigator — Sunway University
Locations (1):
- Department of Psychology, Sunway University, Sunway City, Selangor, Malaysia

REFERENCES:
- [Derived] Ong Lai Teik D, Lee XS, Lim CJ, Low CM, Muslima M, Aquili L. Ginseng and Ginkgo Biloba Effects on Cognition as Modulated by Cardiovascular Reactivity: A Randomised Trial. PLoS One. 2016 Mar 3;11(3):e0150447. doi: 10.1371/journal.pone.0150447. eCollection 2016. PMID 26938637